CLINICAL TRIAL: NCT03977688
Title: Evaluating a CytoSorb Score in Septic Shock - a Retrospective Multicenter Data Analysis
Brief Title: Evaluating a CytoSorb Score in Septic Shock
Acronym: ECSISS
Status: Completed | Type: Observational
Sponsor: Klinikum Emden (Other)
Collaborators: Kantonsspital Münsterlingen (Other); Universitätsklinikum Hamburg-Eppendorf (Other); Kantonsspital Baden (Other)
Responsible Party: Principal Investigator, Klaus Kogelmann, Head of department, Prinipal investigator, Klinikum Emden
Other Study IDs: 20194
Record Dates: First submitted 2019-06-03; First posted 2019-06-06 (Actual); Last update posted 2020-02-19 (Actual); Status verified 2020-02

CONDITIONS: Severe Sepsis With Septic Shock
Keywords: sepsis; septic shock; cytokin adsorption
MeSH Terms: conditions — Sepsis; Shock, Septic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- none Cyto: septic shock, refractory, without Cytokin-adsorption therapy
- cyto: septic shock, refractory, treated with Cytokin-adsorption therapy
  Interventions: Device: Cytokin Adsorption

INTERVENTIONS:
Device: Cytokin Adsorption — Haemadsorption with Cytokin Adsorber (Cytosorb)
  Groups: cyto

SUMMARY:
Systemic hyperinflammatory states, e.g. triggered by infection/sepsis, represent a major challenge for modern medicine. After an initially localized onset, inflammation can extend to an excessive, uncontrolled inflammatory reaction affecting the entire body and can trigger circulatory failure with subsequent irreversible multiple organ failure. Despite all the medical advances made in recent years, sepsis continues to be a substantial problem, as almost all therapeutic approaches have failed to prove their efficacy to date. Mortality in this clinical entity thus remains extremely high. In Germany alone, more than 100,000 people suffer from sepsis or septic shock every year, nearly half of whom die despite optimal therapy. Thus, sepsis is the third most common cause of death, has major importance both from a medical but also from an economical viewpoint, and approaches that could contribute to its successful treatment need to be further developed and explored.

If a patient experiences the spread of bacteria or their constituents in the blood stream due to an uncontrolled source of infection, the result is a deliberately triggered physiological defense reaction of the body. In many patients, however, there is a pathological dysregulation of these mechanisms, in a way that the defense reaction goes far beyond the physiological level required, resulting in an excessive immune response of the body, which is mainly facilitated by inflammatory mediators such as cytokines and chemokines. The immune response spreads throughout the body and also dissipates into organs unaffected by the original infection. In cases of such unwanted overshooting immune responses, an attempt to regain control of the described deleterious systemic events seems reasonable by removing the excess amount of cytokines from the blood, thus preventing or treating organ failure.

In this context, current therapeutic approaches increasingly focus on the elimination of inflammatory mediators.

In recent years, hemoadsorption, using a new adsorber (CytoSorb), has been used to treat sepsis and other conditions of hyperinflammation. The advantage of this therapeutic principle is that a wide range of inflammatory mediators are removed. In conjunction with the enormous elimination capacity, the effective and rapid reduction of mediators can be achieved.

To date, there have been more than 61,000 treatments using this procedure worldwide without device-related side effects being reported. The investigators have been treating patients with this procedure for over 5 years with consistently very favorable results. Therefore, the investigators would like to expand and deepen their observations with the proposed project.

DETAILED DESCRIPTION:
The primary effects of CytoSorb therapy, are, among many others, an improvement in hemodynamics, metobolism, and capillary integrity, with effects of adsorption seeming to reach far beyond mere cytokine adsorption.

Clinically, several publications have shown that certain patient populations benefit most from adjuvant CytoSorb treatment.

In a case series from the investigators department, they examined the effects of CytoSorb as an adjunctive therapy on hemodynamics and on clinically relevant outcome parameters in 26 patients with septic shock and the indication for renal replacement therapy. Treatment was associated with hemodynamic stabilization and reduction in blood lactate levels. The actual mortality was lower than predicted by APACHE II score. This effect was more pronounced in patients in whom therapy was initiated within 24 hours of sepsis diagnosis. Medical patients seemed to benefit more than post-surgical patients in terms of survival.

Based on these results, the investigators performed another study in seven patients with septic shock and ECMO (extracorporeal membrane oxygenation)-dependent acute respiratory distress syndrome (ARDS) treated with a combination therapy of CytoSorb, continuous renal replacement therapy (CRRT) and veno-venous ECMO. The combined treatment was associated with a significant stabilization in hemodynamics and a marked reduction in hyperlactatemia. In addition, patients also showed a significant improvement in lung function and invasiveness of ventilation, and the disease severity and organ dysfunction decreased significantly over the course of the combined treatment, while the observed mortality was only half that predicted by the APACHE II score. The investigators conclude that CytoSorb may be a potentially promising treatment option for patients with refractory ARDS under ECMO therapy in the context of septic shock.

Friesecke et al. prospectively investigated CytoSorb cytokine adsorption in combination with standard of care in 20 patients with refractory septic shock (defined as increasing vasopressor dosages to maintain a MAP of 65mmHg or increasing lactate levels despite protocol-based shock therapy over 6 hours). CytoSorb therapy was started on average after 7.8±3.7 hours of shock therapy. After initiating CytoSorb, norepinephrine dosages could be significantly reduced both after 6 (p=0.03) and 12 (p=0.001) hours. Lactate clearance also improved significantly. Reversal of septic shock was achieved in 13 (65%) patients, with a 28-day survival rate of 45% (with a SOFA predicted mortality of >80%). Treatment with CytoSorb resulted in shock reversal in 2/3 of these difficult-to-treat patients. Data from the CytoSorb registry also support these observations.

In summary, these data show that certain subgroups of patients (in particular those with pneumonia as well as the most critically ill patients with an APACHE score >35) particularly benefit from CytoSorb treatment and that an early onset of therapy (at best <24 hours after diagnosis of septic shock) appears to be beneficial and associated with an increased survival rate.

Given the available information, the investigators analyzed their existing data for dynamic scoring of the first 6 hours in septic shock, based on the study by Ferreira et al. This study showed, that a trend assessment of the SOFA score during the first few days after admission to the intensive care unit allowed for a very good prognosis of the patient's eventual outcome.

The Investigators retrospectively screened data using threshold values for lactate, catecholamine demand, volume requirements, and the need for additional adjuvant therapy with a second catecholamine, and or the application of hydrocortisone.

In this first data analysis, there was an advantage in terms of survival in those patients with pneumonia, in those where Cytosorb therapy was started at least within the first 24 hours of refractory shock, and in patients with slightly higher scores. The investigators subsequently collected this retrospective score in all patients treated at their department who were diagnosed with septic shock according to sepsis-3 criteria in the years 2014-2018. Once again, the benefit - this time also compared to non-Cytosorb-treated patients - could be confirmed.

In order to validate these internal data against neutral other patients, the investigators plan the retrospective data analysis described herein performed as a multi-center study with 3 additional departments which also use CytoSorb therapy. The project involves colleagues from Switzerland (Dr. Hübner, Münsterlingen), Germany (Dr. Jarczak, UK Eppendorf Hamburg) and from Austria (Dr. Schwameis, Baden). Overall, data from approximately 500 patients will be retrospectively collected and analyzed (of which approximately 1/3 patients have been treated with CytoSorb).

The aim is to create a new assessment system based on established, clinically well-available parameters such as lactate, volume and catecholamine therapy to identify patients with early refractory septic shock (Sepsis-3), who would benefit most from adjuvant therapy with Cytosorb hemoadsorption.

For this purpose, physiological patient-related treatment data from patients with septic shock who received CytoSorb treatment will be retrospectively compared to a control group that did not receive this treatment.

Patients who meet the above mentioned inclusion criteria, i.e. who are in a state of septic shock according to the Sepsis-3 definition (sepsis + catecholamine therapy and volume therapy + lactate >2 mmol/l) will be included. Data of included patients will be entered into a data matrix (see chapter 'Assessed parameters'). Each parameter is documented at the time of diagnosis of septic shock as well as 6 hours later to analyze the dynamic process in the early phase of septic shock. The threshold values are based on Sepsis-3 criteria of septic shock (lactate level >2 mmol/l), the administration of norepinephrine according to the SOFA score (norepinephrine > 0.2 μg/kg/min) and volume requirement according to the Surviving Sepsis Guidelines (initial bolus 30 ml/kg body weight).

Each pathological value is rated with 2 points. Decreasing values or no change during the 6 hours observation period receive no points, increasing values receive 1 point, increasing values >50% of the initial value receive 2 points (see data matrix). If <2 volume boluses are necessary, this is rated with 1 point, when ≥2 boluses are necessary within 6 hours, this is scored with 2 points.

In this matrix, septic shock is typically represented by a score of 5 points. Six or more points indicate a situation that is no longer responsive to standard therapy. All data are stored in the respective HIS of the hospitals involved and can be accessed. Centralized data processing will take place at the Department of Anaesthesiology and Intensive Care Medicine at Emden Hospital. The investigators will provide their data anonymously in a tabular format.

Each parameter at the time of septic shock diagnosis (T0h) and 6 hours (T6h) later is documented to analyze the dynamic process in early septic shock.

In addition, values for laboratory diagnostic parameters are also collected 3 days after the diagnosis of septic shock (T72h).

The personal data and findings collected as part of this research project are subject to confidentiality and data protection regulations. They are recorded on paper and stored pseudonymized (encrypted) on data carriers in the participating institutions for a period of 10 years. Name and other identifiers are replaced by a multi-digit code to exclude or substantially complicate the identification of study participants. Only the respective study physician in his or her own center has access to the code which allows a personal assignment of the data of the study participant. As soon as the research purpose allows, the code will be deleted and the data collected will be anonymized. Only the respective study physician can access the data of the patients in their own center. The data are transmitted in a tabular format without any possibility of identification (neither patient-related nor time-related) to the principal study center (Emden Hospital) and provided there with a consecutive number. Access to the data of the individual participating study centers is not possible.

ELIGIBILITY:
Inclusion Criteria:

* septic shock according Sepsis 3 criteria

Exclusion Criteria:

* no data available, no icu treatment

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: each patient eligible with icu treated refractory septic shock in the last 4 years
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Hospital mortality | through study completion, an average of 49 days

SECONDARY OUTCOMES:
Icu mortality | through study completion, an average of 49 days

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Kogelmann, MD, Principal Investigator — head of department
Locations (1):
- Klinikum Emden, Emden, Lower Saxony, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Fleischmann C, Thomas-Rueddel DO, Hartmann M, Hartog CS, Welte T, Heublein S, Dennler U, Reinhart K. Hospital Incidence and Mortality Rates of Sepsis. Dtsch Arztebl Int. 2016 Mar 11;113(10):159-66. doi: 10.3238/arztebl.2016.0159. PMID 27010950
- [Result] Seymour CW, Rosengart MR. Septic Shock: Advances in Diagnosis and Treatment. JAMA. 2015 Aug 18;314(7):708-17. doi: 10.1001/jama.2015.7885. PMID 26284722
- [Result] Iskander KN, Osuchowski MF, Stearns-Kurosawa DJ, Kurosawa S, Stepien D, Valentine C, Remick DG. Sepsis: multiple abnormalities, heterogeneous responses, and evolving understanding. Physiol Rev. 2013 Jul;93(3):1247-88. doi: 10.1152/physrev.00037.2012. PMID 23899564
- [Result] Poli EC, Rimmele T, Schneider AG. Hemoadsorption with CytoSorb(R). Intensive Care Med. 2019 Feb;45(2):236-239. doi: 10.1007/s00134-018-5464-6. Epub 2018 Nov 16. No abstract available. PMID 30446798
- [Result] Kogelmann K, Jarczak D, Scheller M, Druner M. Hemoadsorption by CytoSorb in septic patients: a case series. Crit Care. 2017 Mar 27;21(1):74. doi: 10.1186/s13054-017-1662-9. PMID 28343448
- [Result] Friesecke S, Stecher SS, Gross S, Felix SB, Nierhaus A. Extracorporeal cytokine elimination as rescue therapy in refractory septic shock: a prospective single-center study. J Artif Organs. 2017 Sep;20(3):252-259. doi: 10.1007/s10047-017-0967-4. Epub 2017 Jun 6. PMID 28589286
- [Result] Ferreira FL, Bota DP, Bross A, Melot C, Vincent JL. Serial evaluation of the SOFA score to predict outcome in critically ill patients. JAMA. 2001 Oct 10;286(14):1754-8. doi: 10.1001/jama.286.14.1754. PMID 11594901
- [Result] Singer M, Deutschman CS, Seymour CW, Shankar-Hari M, Annane D, Bauer M, Bellomo R, Bernard GR, Chiche JD, Coopersmith CM, Hotchkiss RS, Levy MM, Marshall JC, Martin GS, Opal SM, Rubenfeld GD, van der Poll T, Vincent JL, Angus DC. The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):801-10. doi: 10.1001/jama.2016.0287. PMID 26903338